CLINICAL TRIAL: NCT00530972
Title: Treatment of Patients With Chronic Hepatitis C Co-infected With HIV Relapsers or Non Responders, Previous Exposed to Sub-optimal Therapies: Open, Pilot Trial
Brief Title: Pilot Study of Patients Chronic Hepatitis C in Co-infected HIV Patients Relapsers After Previous Therapies
Acronym: PILOT-NR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Carlos III, Madrid (Other)
Responsible Party: Vicente Soriano, Hospital Carlos III
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001192-34
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Hepatitis C; HIV Infections
Keywords: co-infected HCV/HIV; relapsers
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peginterferon alfa-2a plus ribavirin (Experimental)
  Interventions: Drug: Peginterferon alfa-2a plus ribavirin adjusted to body weight

INTERVENTIONS:
Drug: Peginterferon alfa-2a plus ribavirin adjusted to body weight — PegInterferon 180 mcg/week, Adjusted body weight Ribavirin (1000 mg <75 kg, 1200 mg >75 kg)

SUMMARY:
To determine the efficacy and safety of Peginterferón alfa-2a (40 KD) plus Ribavirin in patients who have relapsed or not responded to a previous suboptimal therapy based in Interferon.

DETAILED DESCRIPTION:
An important number of co-infected patients were treated suboptimally in the past with others ineffective therapies interferon-based.

All co-infected patients should be an opportunity of retreatment with actually therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 65 years of age
* Anti-HCV positive
* Detectable plasma HCV-RNA
* Relapsers after treatment with interferon o peginterferon +/- ribavirin
* HIV positive
* CD4 >/= 200 cell
* Patients on clinically stable liver disease with:

  * Hgb >/= 12 g/dL in women or 13 g/dL in men
  * Leucocytes >/= 3000 mm3
  * Neutrophil count (ANC) >/= 1500 cells/mm3
  * Platelet count >/= 100.000 cells/mm3
  * Normal prothrombin, bilirubin, albumin, creatinine and uric acid
* HBsAg negative
* With antecedents of diabetes or hypertension is necessary an previous ocular exploration

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, HBeAg
* Hemochromatosis
* Deficit of alfa-1 antitrypsin
* Wilson disease
* Alcoholic liver disease
* Autoimmune hepatitis
* Hepatitis by toxin exposures
* Hepatitis by obesity
* Hemoglobinopathy (e.g. thalassemia)
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Hepatocarcinoma observed in the liver ecography.
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of significant cardiac disease that could be worsened by acute anemia (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina)
* Diabetes Mellitus
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis)
* History or other evidence of chronic pulmonary disease associated with functional limitation
* Drug use within 6 months of 1st dose and excessive alcohol consumption.
* Concomitant treatment with ddI
* Male partners of women who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
% of patients with RNA-HCV undetectable | 24 weeks after end of treatment

SECONDARY OUTCOMES:
% of patients with RNA-HCV undetectable at different moments of the treatment according genotype, viremia, liver fibrosis, number of CD4 cells and previous therapy | At weeks 4, 12, 24 and 48 on treatment
Ribavirin levels | At weeks 4, 12, 24 and 48 on treatment
Impact of dose reduction peg-interferon and/or ribavirin | At weeks 4, 12, 24 and 48 on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Soriano, Dr, Principal Investigator — Hospital Carlos III. Madrid. Spain
Locations (1):
- Hospital Carlos III, Madrid, Madrid, Spain